CLINICAL TRIAL: NCT02647463
Title: Evaluating the Efficacy of ABC for High-Risk Parent and Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Kristin Bernard, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FCNY-73312
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Attachment Disorders
Keywords: Attachment; Cortisol; Parent sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attachment and Biobehavioral Catch-up (Experimental): 10-session intervention for parents and infants aimed at increasing parents' nurturance and following the lead, and reducing frightening behavior
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up (ABC)
- Waitlist Control (No Intervention): Waitlist Control

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-up (ABC)
  Arms: Attachment and Biobehavioral Catch-up

SUMMARY:
Attachment and Biobehavioral Catch-up (ABC) is a manualized 10-session intervention delivered in families' homes or other places of residence. By helping parents of infants provide nurturance when their children are in distress, follow their children's lead, and behave in non-frightening ways, the ABC intervention has been previously found to enhance children's attachment quality and children's ability to regulate behavior, physiology, and emotions. The purpose of the present study is to examine the effectiveness of ABC in the context of community-based implementation efforts. Outcome assessments will include parent sensitivity, attachment quality, and cortisol regulation. The investigators hypothesize that parents randomly assigned to receive the ABC intervention will show higher levels of sensitivity at follow-up than parents randomly assigned to the waitlist control condition; and children randomly assigned to the ABC intervention will show higher rates of secure attachment and more normative profiles of cortisol than children randomly assigned to the waitlist condition.

DETAILED DESCRIPTION:
Chronic stress in early childhood, the result of living in poverty, exposure to violence, and/or experiencing abuse or neglect, undermines a child's development in ways that may have lasting consequences for well-being later in life. High quality parenting (i.e., responding sensitively when children are distressed, and following children's lead) appears to protect against the negative effects of chronic stress, likely by supporting the development of secure attachments and good self-regulation. Unfortunately, many caregivers living in poverty, through no fault of their own, are unable to parent in ways that provide this protection.

Children who face early adversity especially need nurturing, synchronous, and non-frightening care. The ABC intervention was developed to target these three parenting behaviors, with the goal of enhancing attachment relationships and regulatory capacities (Dozier et al., 2011). The ABC intervention is a manualized 10-session program delivered in the parent's home or other place of residence (e.g., homeless shelter). Sessions are videotaped for purposes of video feedback (i.e., showing brief clips back to parents for review of target behaviors), supervision, and fidelity monitoring.

Power of Two is a new non-profit organization in Brooklyn, NY that is implementing the ABC intervention for vulnerable families living in poverty. The purpose of the present study is to examine the effectiveness of ABC in the context of Power of Two's community-based implementation efforts. Using a short-term randomized control design, the investigators aim to replicate and extend previous findings regarding the efficacy of ABC. Participants will include 120 families with infants between 6 months and 20 months of age. Upon referral to the project, families will be randomly assigned to receive the ABC intervention immediately, or be put on a waitlist to receive the ABC intervention after approximately 3 months. Outcome assessments will include: (1) parent sensitivity (assessed at pre-intervention and follow-up), (2) attachment quality (assessed at follow-up), and (3) cortisol regulation (assessed at pre-intervention and follow-up). Additional variables will be included as moderators and covariates.

ELIGIBILITY:
Inclusion Criteria:

* Infant between 6 and 20 months old at time of enrollment
* Living with primary caregiver

Exclusion Criteria:

* Infant will be excluded if he/she has significant medical or developmental problems

Ages: 6 Months to 20 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2016-01; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Attachment organization/security | 1-3 months post-intervention
  Assessed via Strange Situation Procedure (observational)

SECONDARY OUTCOMES:
Diurnal cortisol regulation | 1-3 months post-intervention
  Assessed via saliva samples collected from infants
Parent sensitivity | 1-3 months post-intervention
  Observational assessment of parents' following the lead, intrusiveness, and delight

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bernard, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Power of Two, Brooklyn, New York, United States